CLINICAL TRIAL: NCT00526968
Title: A Double Blind, Placebo Controlled Study to Investigate the Role of NMDA Receptor NR2B Subunit Selective Antagonism on Cognitive Functions and Neurophysiology in Healthy Subjects as Measured With MRI
Brief Title: The Effects of a Novel NMDA NR2B-Subtype Selective Antagonist, EVT 101, on Brain Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Evotec Neurosciences GmbH (Industry)
Collaborators: Richmond Pharmacology Limited (Industry)
Responsible Party: Dr Hermann Fuder, Senior VP, Clinical Development, Evotec Neurosciences GmbH
Organization: Evotec International GmbH (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EVT 101/1002; EudraCT No.: 2007-000986-40
Record Dates: First submitted 2007-09-07; First posted 2007-09-10 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2008-02

CONDITIONS: Human Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): EVT 101 8 mg capsule
  Interventions: Drug: EVT 101
- 2 (Experimental): EVT 101 15 mg capsule
  Interventions: Drug: EVT 101
- 3 (Placebo Comparator): Matching placebo capsule
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: EVT 101 — 8 mg capsule, single oral dose
  Arms: 1
Drug: EVT 101 — 15 mg capsule, single oral dose
  Arms: 2
Drug: placebo — Placebo capsule, single oral dose
  Arms: 3

SUMMARY:
The purpose of this study is to investigate the neurophysiological changes following single doses of EVT 101 using fMRI during rest and during cognitive tasks in young healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male volunteers
* Body Mass Index between 19 and 29

Exclusion Criteria:

* Subjects who received any prescribed medication within 5 half lives or 14 days of the first dose administration whichever is the longer
* Subjects who have received any prescribed CNS medication or any medication known to chronically alter drug absorption or elimination processes within 30 days of first dose administration
* Participation in a clinical trial of an investigational drug within the past 4 months or of a marketed drug within the past 3 months
* History of allergy to NMDA antagonists or other clinically significant drug allergy
* Supine blood pressure and heart rate of higher than 140/90 mmHg and 90 bpm respectively or lower than 80/40 mmHg and 40 bpm
* Consumption of more than 21 units of alcohol per week or history of alcoholism or drug/chemical abuse
* Smokers of more than 5 cigarettes or equivalent per day
* Subjects who cannot complete the neuropsychological test battery
* Any clinically significant health deficit

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Change in fMRI BOLD signal under baseline conditions and during activation by cognitive tasks | 2-hours post dose
Change in regional cerebral blood flow (determined with ASL-MRI)after drug compared with placebo | 2-hours post dose
Performance scores in the cognitive tests | 2-hours post dose

SECONDARY OUTCOMES:
Safety, tolerability, adverse events, safety laboratory tests, ECG, vital signs | Up to 24 hours post dose and 5-7 days post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Leigh, BSc MBBS Phd, Principal Investigator — Department of Clinical Neurosciences, Institute of Psychiatry
Locations (1):
- Centre for Neuroimaging Science, Box 089, Institute of Psychiatry, London, United Kingdom